CLINICAL TRIAL: NCT00882453
Title: Betaferon Treatment and Exercise Data Gathering IN Early MS
Brief Title: Physical Activity and Fatigue in Early Multiple Sclerosis (MS)
Acronym: BEGIN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Regional Medical Director, Bayer Healthcare AG
Other Study IDs: 13853; BF0601 (Other: company internal); 310721 (Other: company internal)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Multiple Sclerosis
Keywords: Physical Activity; Fatigue; RRMS; CIS
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Intravenous therapy according to product information

SUMMARY:
The purpose of this observational study is to obtain a survey on physical activity in patients who for the first time have experienced symptoms which indicate a high risk for developing multiple sclerosis (MS) and in patients with recently diagnosed MS, and to obtain information on factors potentially influencing the patients' level of activity.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis diagnosed within the last 12 months
* Clinically isolated Syndrome (CIS), under Interferon-beta-1b treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after a first demyelinating event suggestive of MS as well as patients with recently diagnosed RRMS (< 12 months)
Sampling Method: Non-Probability Sample
Enrollment: 1739 (Actual)
Dates: Start 2006-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Physical Activity and Fatigue | At baseline and at Month 24

SECONDARY OUTCOMES:
Health-related Quality of Life | At baseline and at Month 24
Depression | At baseline and at Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Many Locations, Australia
- Many Locations, Austria
- Many Locations, Bahrain
- Many Locations, Belgium
- Many Locations, Canada
- Many Locations, Colombia
- Many Locations, Czechia
- Many Locations, Denmark
- Many Locations, Egypt
- Many Locations, France
- Many Locations, Germany
- Many Locations, Greece
- Many Locations, Indonesia
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Jordan
- Many Locations, Kazakhstan
- Many Locations, Kuwait
- Many Locations, Lebanon
- Many Locations, Mexico
- Many Locations, Netherlands
- Many Locations, Norway
- Many Locations, Oman
- Many Locations, Portugal
- Many Locations, Slovenia
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Switzerland
- Many Locations, Taiwan
- Many Locations, Thailand
- Many Locations, United Arab Emirates
- Many Locations, United Kingdom